CLINICAL TRIAL: NCT00194064
Title: Pilot Study Evaluating the Safety and Efficacy of Open-Label Olanzapine Monotherapy in Treatment Refractory Bipolar Disorder Mania
Brief Title: Pilot Study Evaluating the Safety and Efficacy of Open-Label Olanzapine
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Joseph Calabrese, MD, Director, Mood Disorders Program, University Hospitals Cleveland Medical Center
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F1DMC-X136
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olanzapine (Experimental): Subjects were be started on a standardized minimum first-day dose of 15 mg olanzapine. After the first day of therapy, the daily dose was either increased or decreased, as clinically indicated, by 5 mg, within an allowed range of 5 to 40 mg
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine
  Other Names: Zyprexa

SUMMARY:
Inpatient Study Evaluating the Safety and Efficacy of Open-Label Olanzapine Monotherapy in Treatment Refractory Bipolar Mania: This study recruits adult subjects who are diagnosed with Bipolar I Disorder and presently experiencing an episode of mania. Patients must be willing to spend initial 7 days in the hospital to observe response to medication. Patients must be refractory (intolerant or non-responsive) to treatment with lithium and valproate or carbamazepine. Patients receive study-related care at no cost. This study is sponsored by Eli Lilly and Company.

ELIGIBILITY:
Inclusion Criteria:

* The subject satisfied Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for a primary diagnosis of Bipolar Disorder, most recently manic
* The patient is willing to be hospitalized on an inpatient psychiatric unit for a minimum of seven (7) days.
* Subject has been treated with lithium in the past.
* Subject has been treated with divalproex or carbamazepine in the past.
* Subject has been treated with Haldol or haloperidol in the past.

Exclusion Criteria:

* Subjects lacks the capacity to provide informed consent
* Subject is a serious suicide risk or has medically unstable conditions as judged by the investigators
* Subject has been dependent on a drug (other than nicotine or caffeine) in the last three (3) months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-07; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale (YMRS) | Change from Baseline to End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Calabrese, MD, Principal Investigator — Case Western Reserve University / University Hospitals of Cleveland
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States